CLINICAL TRIAL: NCT04228237
Title: LUng CAncer focuS - Long Term Non-interventional Monitoring of Diagnostic and Treatment Patterns in Patients With Bronchogenic Carcinoma (LUCAS)
Brief Title: LUng CAncer focuS - Long-term Monitoring of Bronchogenic Carcinoma Patients (LUCAS)
Acronym: LUCAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ceska Lekarska Spolecnost Jana Evangelisty Purkyne z.s. (Other)
Collaborators: OAKS Consulting s.r.o. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CPFS/Reg18.01
Record Dates: First submitted 2019-10-31; First posted 2020-01-14 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
Keywords: lung cancer; bronchogenic carcinoma; diagnosis; treatment; non-interventional
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Bronchogenic; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term non-interventional monitoring of diagnostics and treatment patterns in newly diagnosed patients in selected pneumology centers in Czech republic.

DETAILED DESCRIPTION:
Diagnosis, treatment and care of patients with bronchogenic carcinoma (BCA) is, as with most other oncological diseases, a complex multidisciplinary process. Due to the lack of information on the speed and success of the initial diagnosis, the use of the necessary laboratory techniques, and the individual therapeutic steps leading to cure or medical failure, the Czech Pneumological and Phtizeology Society (CPPS) decided to carry out long-term non-interventional monitoring of newly diagnosed patients.

This monitoring is non-interventional, so the usual diagnostic and therapeutic procedures will be used according to the decision of the physician. All patients with bronchogenic carcinoma diagnosed from June 1, 2018 will be enrolled with up to 60 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

- clinical diagnosis of lung cancer (C34 in MKN classification)

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all newly diagnosed patients in participating pulmonology centers
Sampling Method: Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 60 months of follow-up
  Time from randomization until death from any cause
Progression-free survival (PFS) | any treatment during 60 months of follow-up
  Time from randomization until disease progression or death
Time to treatment discontinuation (TTD) | any treatment during 60 months of follow-up
  time from starting a medication until treatment discontinuation or death

SECONDARY OUTCOMES:
Time to next treatment (TTNT) | 60 months of follow-up
  Time from end of primary treatment to institution of next therapy

CONTACTS AND LOCATIONS:
Overall Officials: Martina Koziar Vasakova, Prof., Principal Investigator — University Thomayer hospital Prague
Locations (7):
- Czechia (7):
  - University hospital Brno, Brno
  - University hospital Hradec Kralove, Hradec Králové
  - University hospital Olomouc, Olomouc
  - University hospital Plzen, Pilsen
  - University Thomayer hospital, Prague
  - University hospital Motol, Prague
  - University hospital Bulovka, Prague, Česká Republika

REFERENCES:
- [Derived] Venclicek O, Skrickova J, Brat K, Fischer O, Havel L, Hrnciarik M, Marel M, Opalka P, Krakorova G, Rozsivalova D, Kultan J, Mullerova A, Zarnayova L, Smickova P, Vasakova M, Gyorfy Z, Jirousek M, Krejci D, Krejci J, Zuna P, Svaton M, Hrda K, Duba J, Alahakoon J, Svoboda M, Silar J. Lung Cancer in Non-smokers in Czech Republic: Data from LUCAS Lung Cancer Clinical Registry. Anticancer Res. 2021 Nov;41(11):5549-5556. doi: 10.21873/anticanres.15368. PMID 34732425